CLINICAL TRIAL: NCT00950118
Title: Diaphragmatic Hernia Research & Exploration, Advancing Molecular Science
Acronym: DHREAMS
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAB2063; R01HD057036 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Congenital Diaphragmatic Hernia (CDH); Genes; Genetic; Genetic testing; exome sequencing; genome sequencing; RNAseq
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, tissue, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenital Diaphragmatic Hernia (CDH): Humans affected with congenital diaphragmatic hernia (CDH)
- Unaffected: Healthy family members of individuals affected with congenital diaphragmatic hernia (CDH)

SUMMARY:
The goal of this study is to identify genes that convey susceptibility to congenital diaphragmatic hernia in humans. The identification of such genes, and examination of their structure and function, will enable a delineation of molecular pathogenesis and, ultimately, prevention or treatment of congenital diaphragmatic hernia. There are many different possible modes of inheritance for congenital anomalies, including autosomal dominant, autosomal recessive, and multifactorial. Multi-factorial inheritance is responsible for many common medical disorders, including hypertension, myocardial infarction, diabetes and cancer. This type of inheritance pattern appears to involve environmental factors as well as a combination of genetic variations that together can predispose to or produce congenital anomalies, such as congenital diaphragmatic hernia.

Our study is designed to establish a small, well-defined genetic resource consisting of 1) Nuclear families suitable for linkage analysis by parametric,non-parametric (e.g. sib pairs, TDT) and association techniques, 2) Individuals with congenital diaphragmatic hernia who can be directly screened for allelic variation in candidate genes, and 3) Individuals who can serve as controls (are unaffected by congenital diaphragmatic hernia). Neonates and their families will be collected from homogenous and heterogeneous populations. By characterizing diverse populations, it should be possible to increase the likelihood of demonstration of genetic variation in selected candidate genes that can then be used in association and linkage studies in individual subjects with congenital diaphragmatic hernia.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a birth defect that occurs when the diaphragm (thin sheet of muscle that separates the abdomen from the chest) does not form properly. When an opening is present in the diaphragm, organs that are normally in the abdomen can be pushed (herniated) through the opening and be present in the chest. Currently little is known about why this birth defect occurs.

Through this study ""Molecular Genetic Analysis of Congenital Diaphragmatic Hernia" the investigators hope to learn more about whether certain genes contribute to CDH. Genes are the instructions or blueprints for our bodies. They tell our bodies how to grow and develop. Sometimes when a mistake occurs in one or more of our genes our body does not develop properly and this can lead to a CDH. The investigators hope that the information gained through studying the genes of children with CDH and their parents, will lead to significant advances in the diagnosis, prognosis, prevention, and treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* All individuals affected with a congenital diaphragmatic hernia (CDH), or with a family history of a CDH

Exclusion Criteria:

* Individuals with no personal history of a CDH or family history of a family member affected with congenital diaphragmatic hernia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children/neonates with an unrepaired congenital diaphragmatic hernia
  Children/neonates with a reparied congenital diaphragmatic hernia
  Women who are pregnant with a fetus diagnosed with congenital diaphragmatic hernia
  Individuals with a family history of congenital diaphragmatic hernia
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2005-06; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a genetic diagnosis | 5 years
  DNA samples from patients will be analyzed for underlying genetic causes.

SECONDARY OUTCOMES:
Developmental outcomes at 2 and 5 years of age | 1 exam at 2 year and 1 exam at 5 years
  Formal Developmental outcome measures
Percentage of patients with pulmonary hypertension | 5 years
  pulmonary hypertension measured by echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Shen, PhD, Principal Investigator — Columbia University
Locations (14):
- United States (13):
  - Rush Hospital, Chicago, Illinois
  - University of Michigan/ CS Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University Medical Center/ St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha/ University of Nebraska, Omaha, Nebraska
  - Northwell Health, Manhasset, New York
  - New York University, Hassenfeld Children's Hospital at NYU Langone Health, New York, New York
  - Morgan Stanley Children's Hospital of New York- Presbyterian (Columbia University Medical Center), New York, New York
  - Cincinnati Children's Hospital and Medical Center/ University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Pittsburgh/ University of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carrell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - UT Southwestern Medical Center, Children's Health, Dallas, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wynn J, Yu L, Chung WK. Genetic causes of congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2014 Dec;19(6):324-30. doi: 10.1016/j.siny.2014.09.003. Epub 2014 Oct 28. PMID 25447988
- [Background] Pierog A, Aspelund G, Farkouh-Karoleski C, Wu M, Kriger J, Wynn J, Krishnan U, Mencin A. Predictors of low weight and tube feedings in children with congenital diaphragmatic hernia at 1 year of age. J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):527-30. doi: 10.1097/MPG.0000000000000454. PMID 24918983
- [Background] Yu L, Bennett JT, Wynn J, Carvill GL, Cheung YH, Shen Y, Mychaliska GB, Azarow KS, Crombleholme TM, Chung DH, Potoka D, Warner BW, Bucher B, Lim FY, Pietsch J, Stolar C, Aspelund G, Arkovitz MS; University of Washington Center for Mendelian Genomics; Mefford H, Chung WK. Whole exome sequencing identifies de novo mutations in GATA6 associated with congenital diaphragmatic hernia. J Med Genet. 2014 Mar;51(3):197-202. doi: 10.1136/jmedgenet-2013-101989. Epub 2014 Jan 2. PMID 24385578
- [Background] Wynn J, Aspelund G, Zygmunt A, Stolar CJ, Mychaliska G, Butcher J, Lim FY, Gratton T, Potoka D, Brennan K, Azarow K, Jackson B, Needelman H, Crombleholme T, Zhang Y, Duong J, Arkovitz MS, Chung WK, Farkouh C. Developmental outcomes of children with congenital diaphragmatic hernia: a multicenter prospective study. J Pediatr Surg. 2013 Oct;48(10):1995-2004. doi: 10.1016/j.jpedsurg.2013.02.041. PMID 24094947
- [Background] Wynn J, Krishnan U, Aspelund G, Zhang Y, Duong J, Stolar CJ, Hahn E, Pietsch J, Chung D, Moore D, Austin E, Mychaliska G, Gajarski R, Foong YL, Michelfelder E, Potolka D, Bucher B, Warner B, Grady M, Azarow K, Fletcher SE, Kutty S, Delaney J, Crombleholme T, Rosenzweig E, Chung W, Arkovitz MS. Outcomes of congenital diaphragmatic hernia in the modern era of management. J Pediatr. 2013 Jul;163(1):114-9.e1. doi: 10.1016/j.jpeds.2012.12.036. Epub 2013 Jan 30. PMID 23375362
- [Background] Yu L, Wynn J, Cheung YH, Shen Y, Mychaliska GB, Crombleholme TM, Azarow KS, Lim FY, Chung DH, Potoka D, Warner BW, Bucher B, Stolar C, Aspelund G, Arkovitz MS, Chung WK. Variants in GATA4 are a rare cause of familial and sporadic congenital diaphragmatic hernia. Hum Genet. 2013 Mar;132(3):285-92. doi: 10.1007/s00439-012-1249-0. Epub 2012 Nov 9. PMID 23138528
- [Background] Yu L, Wynn J, Ma L, Guha S, Mychaliska GB, Crombleholme TM, Azarow KS, Lim FY, Chung DH, Potoka D, Warner BW, Bucher B, LeDuc CA, Costa K, Stolar C, Aspelund G, Arkovitz MS, Chung WK. De novo copy number variants are associated with congenital diaphragmatic hernia. J Med Genet. 2012 Oct;49(10):650-9. doi: 10.1136/jmedgenet-2012-101135. PMID 23054247
- [Background] Yu L, Sawle AD, Wynn J, Aspelund G, Stolar CJ, Arkovitz MS, Potoka D, Azarow KS, Mychaliska GB, Shen Y, Chung WK. Increased burden of de novo predicted deleterious variants in complex congenital diaphragmatic hernia. Hum Mol Genet. 2015 Aug 15;24(16):4764-73. doi: 10.1093/hmg/ddv196. Epub 2015 Jun 1. PMID 26034137
- [Background] Azarow KS, Cusick R, Wynn J, Chung W, Mychaliska GB, Crombleholme TM, Chung DH, Lim FY, Potoka D, Warner BW, Aspelund G, Arkovitz MS. The association between congenital diaphragmatic hernia and undescended testes. J Pediatr Surg. 2015 May;50(5):744-5. doi: 10.1016/j.jpedsurg.2015.02.025. Epub 2015 Feb 19. PMID 25783379
- [Background] Kardon G, Ackerman KG, McCulley DJ, Shen Y, Wynn J, Shang L, Bogenschutz E, Sun X, Chung WK. Congenital diaphragmatic hernias: from genes to mechanisms to therapies. Dis Model Mech. 2017 Aug 1;10(8):955-970. doi: 10.1242/dmm.028365. PMID 28768736
- [Background] Kruszka P, Tanpaiboon P, Neas K, Crosby K, Berger SI, Martinez AF, Addissie YA, Pongprot Y, Sittiwangkul R, Silvilairat S, Makonkawkeyoon K, Yu L, Wynn J, Bennett JT, Mefford HC, Reynolds WT, Liu X, Mommersteeg MTM, Chung WK, Lo CW, Muenke M. Loss of function in ROBO1 is associated with tetralogy of Fallot and septal defects. J Med Genet. 2017 Dec;54(12):825-829. doi: 10.1136/jmedgenet-2017-104611. Epub 2017 Jun 7. PMID 28592524
- [Background] Longoni M, High FA, Qi H, Joy MP, Hila R, Coletti CM, Wynn J, Loscertales M, Shan L, Bult CJ, Wilson JM, Shen Y, Chung WK, Donahoe PK. Genome-wide enrichment of damaging de novo variants in patients with isolated and complex congenital diaphragmatic hernia. Hum Genet. 2017 Jun;136(6):679-691. doi: 10.1007/s00439-017-1774-y. Epub 2017 Mar 16. PMID 28303347
- [Background] Chiu JS, Ma L, Wynn J, Krishnan U, Rosenzweig EB, Aspelund G, Arkovitz M, Warner BW, Lim FY, Mychaliska GB, Azarow K, Cusick RA, Chung DH, Chung WK. Mutations in BMPR2 are not present in patients with pulmonary hypertension associated with congenital diaphragmatic hernia. J Pediatr Surg. 2017 Nov;52(11):1747-1750. doi: 10.1016/j.jpedsurg.2017.01.007. Epub 2017 Jan 26. PMID 28162765
- [Background] Farkouh-Karoleski C, Najaf T, Wynn J, Aspelund G, Chung WK, Stolar CJ, Mychaliska GB, Warner BW, Wagner AJ, Cusick RA, Lim FY, Schindel DT, Potoka D, Azarow K, Cotten CM, Hesketh A, Soffer S, Crombleholme T, Needelman H. A definition of gentle ventilation in congenital diaphragmatic hernia: a survey of neonatologists and pediatric surgeons. J Perinat Med. 2017 Dec 20;45(9):1031-1038. doi: 10.1515/jpm-2016-0271. PMID 28130958
- [Background] Abramov A, Fan W, Hernan R, Zenilman AL, Wynn J, Aspelund G, Khlevner J, Krishnan U, Lim FY, Mychaliska GB, Warner BW, Cusick R, Crombleholme T, Chung D, Danko ME, Wagner AJ, Azarow K, Schindel D, Potoka D, Soffer S, Fisher J, McCulley D, Farkouh-Karoleski C, Chung WK, Duron V. Comparative outcomes of right versus left congenital diaphragmatic hernia: A multicenter analysis. J Pediatr Surg. 2020 Jan;55(1):33-38. doi: 10.1016/j.jpedsurg.2019.09.046. Epub 2019 Oct 26. PMID 31677822
- [Background] Qiao L, Wynn J, Yu L, Hernan R, Zhou X, Duron V, Aspelund G, Farkouh-Karoleski C, Zygumunt A, Krishnan US, Nees S, Khlevner J, Lim FY, Crombleholme T, Cusick R, Azarow K, Danko ME, Chung D, Warner BW, Mychaliska GB, Potoka D, Wagner AJ, Soffer S, Schindel D, McCulley DJ, Shen Y, Chung WK. Likely damaging de novo variants in congenital diaphragmatic hernia patients are associated with worse clinical outcomes. Genet Med. 2020 Dec;22(12):2020-2028. doi: 10.1038/s41436-020-0908-0. Epub 2020 Jul 28. PMID 32719394
- [Background] Yu L, Hernan RR, Wynn J, Chung WK. The influence of genetics in congenital diaphragmatic hernia. Semin Perinatol. 2020 Feb;44(1):151169. doi: 10.1053/j.semperi.2019.07.008. Epub 2019 Aug 1. PMID 31443905
- See also: Study Website — http://www.cdhgenetics.com